CLINICAL TRIAL: NCT02443493
Title: Low-level Laser Therapy as a Tool for the Prevention of Radiodermatitis in Breast Cancer Patients
Brief Title: Laser Therapy for the Prevention of Radiodermatitis in Breast Cancer Patients
Acronym: TRANSDERMIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Collaborators: Jessa Hospital (Other)
Responsible Party: Principal Investigator, Prof. dr. Jeroen Mebis, prof. dr., Hasselt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 15.38/onco15.06
Record Dates: First submitted 2015-05-11; First posted 2015-05-13 (Estimated); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Low-Level Light Therapy; Radiotherapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment group (Experimental): Treatment group (receives low-level laser therapy (2x/week) in combination with standard skin care starting from day 1 of radiotherapy)
  Interventions: Device: Low-level laser; Radiation: radiotherapy
- Control group (Sham Comparator): Control group (receives sham laser (2x/week) in combination with standard skin care starting from day 1 of radiotherapy)
  Interventions: Device: sham laser; Radiation: radiotherapy

INTERVENTIONS:
Device: Low-level laser — Low-Level Laser Therapy will be applied, twice a week, from the start of radiotherapy treatment (14 sessions in total) in combination with the standard skin care.
  Other Names: LLLT
  Arms: Treatment group
Device: sham laser — Sham Laser Therapy will be applied, twice a week, from the start of radiotherapy treatment (14 sessions in total) in combination with the standard skin care.
  Arms: Control group
Radiation: radiotherapy

SUMMARY:
Up to 90% of the radiotherapy patients will develop a certain degree of skin reaction at the treated area, also known as radiodermatitis (RD).

Currently, there is a wide variety of strategies to manage RD, including creams, gels, ointments, wound dressings. However, up to now, there is still no comprehensive, evidence-based consensus for the treatment of RD. Low-level laser therapy (LLLT) is a promising, non-invasive technique for treating RD. In a recent pilot study conducted in our research group, LLLT prevented the aggravation of RD and provided symptomatic relief in patients undergoing radiotherapy for breast cancer after breast-sparing surgery. This pilot study was the first prospective study investigating the potential of LLLT for RD. In the current study, we want to investigate the efficacy of LLLT as a tool for the prevention of radiodermatitis in breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of non-invasive (stage 0) or invasive (stage 1, 2 and 3A) breast adenocarcinoma
* Treatment with primary breast-sparing surgery (lumpectomy) and/or neoadjuvant (preoperative) or adjuvant (postoperative) chemotherapy or hormonal therapy
* Scheduled for postoperative radiotherapy with standard technique (isocentric) and fractionation regime (i.e. 25 daily fractions of 2 Gray to the whole breast followed by a boost of 8 fractions of 2 Gray to the tumor bed, 5/week)
* Signed informed consent

Exclusion Criteria:

* Previous irradiation to the same breast
* Metastatic disease
* Concurrent chemotherapy
* Required use of bolus material to deliver radiotherapy (i.e. material placed on the to- be-irradiated zone to modulate the delivered dose in order the ensure an optimal distribution of the radiation dose; mostly used for treatment of superficial tumors)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Radiation Dermatitis Grade | day 1
  objective scoring of the severity of radiation dermatitis using the grading system of the Radiation Therapy Oncology Group/ European Organization for Research and Treatment of Cancer (RTOG/ EORTC)
Radiation Dermatitis Grade | day 20
  objective scoring of the severity of radiation dermatitis using the grading system of the Radiation Therapy Oncology Group/ European Organization for Research and Treatment of Cancer (RTOG/ EORTC)
Radiation Dermatitis Grade | day 33
  objective scoring of the severity of radiation dermatitis using the grading system of the Radiation Therapy Oncology Group/ European Organization for Research and Treatment of Cancer (RTOG/ EORTC)
Radiation Dermatitis Grade | day 40
  objective scoring of the severity of radiation dermatitis using the grading system of the Radiation Therapy Oncology Group/ European Organization for Research and Treatment of Cancer (RTOG/ EORTC)
Radiation Dermatitis Grade | day 54
  objective scoring of the severity of radiation dermatitis using the grading system of the Radiation Therapy Oncology Group/ European Organization for Research and Treatment of Cancer (RTOG/ EORTC)
Radiation Dermatitis Assessment | day 1
  radiation dermatitis assessment scale (Radiation-Induced Skin Reaction Assessment Scale, RISRAS)
Radiation Dermatitis Assessment | day 20
  radiation dermatitis assessment scale (Radiation-Induced Skin Reaction Assessment Scale, RISRAS)
Radiation Dermatitis Assessment | day 33
  radiation dermatitis assessment scale (Radiation-Induced Skin Reaction Assessment Scale, RISRAS)
Radiation Dermatitis Assessment | day 40
  radiation dermatitis assessment scale (Radiation-Induced Skin Reaction Assessment Scale, RISRAS)
Radiation Dermatitis Assessment | day 54
  radiation dermatitis assessment scale (Radiation-Induced Skin Reaction Assessment Scale, RISRAS)
Objective measurement of trans epidermal water loss of the skin | day 1
  Tewa meter TM 300 will be used to objectively assess the skin barrier function by measuring the trans epidermal water loss of the skin
Objective measurement of trans epidermal water loss of the skin | day 20
  Tewa meter TM 300 will be used to objectively assess the skin barrier function by measuring the trans epidermal water loss of the skin
Objective measurement of trans epidermal water loss of the skin | day 33
  Tewa meter TM 300 will be used to objectively assess the skin barrier function by measuring the trans epidermal water loss of the skin
Objective measurement of trans epidermal water loss of the skin | day 40
  Tewa meter TM 300 will be used to objectively assess the skin barrier function by measuring the trans epidermal water loss of the skin
Objective measurement of trans epidermal water loss of the skin | day 54
  Tewa meter TM 300 will be used to objectively assess the skin barrier function by measuring the trans epidermal water loss of the skin
Objective measurement of the skin hydration | day 1
  Corneo meter CM825 will be used to objectively assess the skin barrier function by measuring the skin hydration
Objective measurement of the skin hydration | day 20
  Corneo meter CM825 will be used to objectively assess the skin barrier function by measuring the skin hydration
Objective measurement of the skin hydration | day 33
  Corneo meter CM825 will be used to objectively assess the skin barrier function by measuring the skin hydration
Objective measurement of the skin hydration | day 40
  Corneo meter CM825 will be used to objectively assess the skin barrier function by measuring the skin hydration
Objective measurement of trans epidermal water loss of the skin | day 54
  Corneo meter CM825 will be used to objectively assess the skin barrier function by measuring the skin hydration
Objective measurement of degree of erythema of the skin | day 1
  Mexa meter MX18 will be used to objectively measure the degree of erythema of the skin
Objective measurement of degree of erythema of the skin | day 20
  Mexa meter MX18 will be used to objectively measure the degree of erythema of the skin
Objective measurement of degree of erythema of the skin | day 33
  Mexa meter MX18 will be used to objectively measure the degree of erythema of the skin
Objective measurement of degree of erythema of the skin | day 40
  Mexa meter MX18 will be used to objectively measure the degree of erythema of the skin
Objective measurement of degree of erythema of the skin | day 54
  Mexa meter MX18 will be used to objectively measure the degree of erythema of the skin
Analyze the skin cytokine content of the irradiated and non-irradiated breast | day 1
  Collect skin tape samples of the irradiated and non-irradiated breast in order to analyze these samples on cytokines by ELISA
Analyze the skin cytokine content of the irradiated and non-irradiated breast | day 20
  Collect skin tape samples of the irradiated and non-irradiated breast in order to analyze these samples on cytokines by ELISA
Analyze the skin cytokine content of the irradiated and non-irradiated breast | day 33
  Collect skin tape samples of the irradiated and non-irradiated breast in order to analyze these samples on cytokines by ELISA
Analyze the skin cytokine content of the irradiated and non-irradiated breast | day 40
  Collect skin tape samples of the irradiated and non-irradiated breast in order to analyze these samples on cytokines by ELISA
Analyze the skin cytokine content of the irradiated and non-irradiated breast | day 54
  Collect skin tape samples of the irradiated and non-irradiated breast in order to analyze these samples on cytokines by ELISA

SECONDARY OUTCOMES:
Pain | day 1
  Evaluation of pain using a Visual Analogue Scale (VAS)
Pain | day 20
  Evaluation of pain using a Visual Analogue Scale (VAS)
Pain | day 33
  Evaluation of pain using a Visual Analogue Scale (VAS)
Pain | day 40
  Evaluation of pain using a Visual Analogue Scale (VAS)
Pain | day 54
  Evaluation of pain using a Visual Analogue Scale (VAS)
Quality of life | day 1
  Health-related quality of life measure specific to skin diseases
Quality of life | day 20
  Health-related quality of life measure specific to skin diseases
Quality of life | day 33
  Health-related quality of life measure specific to skin diseases
Quality of life | day 40
  Health-related quality of life measure specific to skin diseases
Quality of life | day 54
  Health-related quality of life measure specific to skin diseases
Satisfaction with therapy | day 1
  Self-report on the efficacy of and the global satisfaction with the management of radiodermatitis
Satisfaction with therapy | day 20
  Self-report on the efficacy of and the global satisfaction with the management of radiodermatitis
Satisfaction with therapy | day 33
  Self-report on the efficacy of and the global satisfaction with the management of radiodermatitis
Satisfaction with therapy | day 40
  Self-report on the efficacy of and the global satisfaction with the management of radiodermatitis
Satisfaction with therapy | day 54
  Self-report on the efficacy of and the global satisfaction with the management of radiodermatitis
moist desquamation | day 1
  3 months (during radiotherapy + 1 month after radiotherapy) Description: Onset time of moist desquamation
moist desquamation | day 20
  3 months (during radiotherapy + 1 month after radiotherapy) Description: Onset time of moist desquamation
moist desquamation | day 33
  3 months (during radiotherapy + 1 month after radiotherapy) Description: Onset time of moist desquamation
moist desquamation | day 40
  3 months (during radiotherapy + 1 month after radiotherapy) Description: Onset time of moist desquamation
moist desquamation | day 54
  3 months (during radiotherapy + 1 month after radiotherapy) Description: Onset time of moist desquamation

CONTACTS AND LOCATIONS:
Overall Officials: Jeroen Mebis, prof. dr., Principal Investigator — Universiteit Hasselt/ Jessa ziekenhuis
Locations (1):
- Jessa Hospital - Oncology department, Hasselt, Belgium